CLINICAL TRIAL: NCT03225456
Title: Exploring the Effects of Oxytocin on Appetite Regulation in Healthy Adult Men
Brief Title: Oxytocin and Eating
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yale-NUS College (Other)
Collaborators: Singapore General Hospital (Other); SingHealth Investigational Medicine Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IG15-LR052
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Weight Gain
Keywords: appetite regulation; obesity; oxytocin
MeSH Terms: conditions — Weight Gain; Obesity | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Participants will receive two doses of 24 IU intra-nasal oxytocin (Syntocinon) in a single session
  Interventions: Drug: Syntocinon
- Placebo (Placebo Comparator): Participants will received match placebo, again in two doses in a single session
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Syntocinon — Intra-nasal oxytocin
  Arms: Oxytocin
Drug: Placebos — Intra-nasal placebo
  Arms: Placebo

SUMMARY:
In this protocol, the investigators propose a randomised controlled trial to explore the effects of intra-nasal oxytocin administration on appetite regulation. The investigators will run a cross-over design with 60 healthy adult men.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Age: 21-45 years
* Normal weight: Body mass index of 18.5 to 22.9
* Have had a stable weight for the past 3 months (less than 5kg)
* Have regular breakfast meals (≥ 4 times a week of self-reported consumption of a breakfast meal)
* Have habitual sleep of 6.5-8.5 hours
* Have English as first language (or fluent in spoken and written English)

Exclusion Criteria:

* Symptoms / history of any major medical condition, including:

  * Bariatric surgery or surgical obesity treatment
  * Diabetes
  * Cardiovascular disease
  * Thyroid disease
  * Anaemia
  * Psychiatric disorders
  * Eating disorders
* Excessive exercise (running > 40 km or exercising > 10 hr in a week)
* Currently on a special diet or trying deliberately to restrict food intake
* Currently on a weight loss program
* Smoking or substance abuse
* Use of medications that can affect weight (e.g., steroids, approved weight-loss drugs)

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Taste sensitivity | 2-hour span following oxytocin administration
  Taste thresholds for primary taste senses, measured using psychophysical staircase procedures
Taste preference | 2-hour span following oxytocin administration
  Measured using the positive/negative generalised Labeled Magnitude Scale used to
  assess pleasantness
Value placed upon food | 2-hour span following oxytocin administration
  Willingness to pay for food (vs non-food items) in a Becker-DeGroot-Marschak auction task

SECONDARY OUTCOMES:
Subjective ratings of hunger and fullness | 2-hour span following oxytocin administration
  Measured using 100-point Visual Analogue Scales

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No